CLINICAL TRIAL: NCT00149526
Title: Does Shared Decision-Making Improve Asthma Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 261; R01HL067092 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: Shared Decision-Making

SUMMARY:
To improve asthma outcomes by developing and evaluating strategies for enhancing the clinic-patient partnership. To develop a model of shared decision-making for asthma treatment, and to evaluate it in a two-year randomized clinical trial in 342 adults aged 18-70 years with sub-optimally controlled persistent asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Although much is now known about asthma, and there is effective asthma treatment, only about half of the patients with persistent asthma adhere to their prescribed long-term controller medication. One way to change this might be to involve patients more in decisions about their treatment.

DESIGN NARRATIVE:

Overview and study design This study is designed to evaluate the effectiveness of a model of shared decision-making in improving outcomes in adults aged 18-70 years with suboptimally controlled, mild-moderate persistent asthma. The shared decision-making model (SD) is being compared in a randomized controlled trial with a model based on national asthma guidelines (MG), and with usual care (UC).

Initially, we adapted the model of shared decision-making that has been used successfully in cancer to make it appropriate for a chronic disease (asthma). We will also adapted the KP Asthma Guidelines so that the two models (Management by Guidelines and Shared Decision-Making) take a similar amount of clinician-patient interaction time. We are comparing the two models and usual care in the primary care setting at Kaiser Permanente Northwest and Kaiser Permanente Hawaii in a randomized controlled trial with 24-month follow up. The individual asthma patient will be the unit of randomization.

Interventions were done by a care manager (nurse practitioner or clinical pharmacist) with experience in asthma, and the authority to change medication regimens. Different staff were used for the two intervention groups to minimize contamination between the groups attributable to the intervention. Eligible participants were randomized into the three groups (UC, MG, and SD) on an equal 1:1:1 basis, stratifying on prior health care utilization and within center (KPNW or KPH). All study participants are being followed for 24 months with clinic visits for data collection at 12 months. The MG and SD arms are receiving interim phone calls from the care managers at three, six, and nine months to assess problems with their treatment regimens, discuss changes that may be desired in treatment regimens, and encourage adherence. Different staff are responsible for data collection and intervention.

We will compare the MG and SD models versus usual care (UC vs MG; UC vs SD), and the MG and SD models (MG vs SD).

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Inclusion: Asthma not well-controlled; doctor-diagnosed asthma; currently taking asthma medications; 12 % and 200ml increase in FEV1 after 2 puffs of an inhaled short-acting -agonist (SABA) bronchodilator ; 2 or more control problems identified using the ATAQ asthma control instrument; 18-70 years of age; willing to be randomized to one of the three treatment arms and to participate in follow-up for 2 years; Kaiser Permanente member for 1 year

Exclusion: Mild intermittent asthma, defined as either seasonal asthma or (daytime asthma symptoms <2x/week and nocturnal symptoms <2x/month and no use of controller medications); under the ongoing care of an allergist or pulmonologist; regular use of oral corticosteroids; currently receiving case-management for their asthma; unable to speak, read or understand English; planning to leave the catchment area within the next two years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Study Completion 2006-05 (Actual)

REFERENCES:
- [Derived] Wilson SR, Strub P, Buist AS, Knowles SB, Lavori PW, Lapidus J, Vollmer WM; Better Outcomes of Asthma Treatment (BOAT) Study Group. Shared treatment decision making improves adherence and outcomes in poorly controlled asthma. Am J Respir Crit Care Med. 2010 Mar 15;181(6):566-77. doi: 10.1164/rccm.200906-0907OC. Epub 2009 Dec 17. PMID 20019345